CLINICAL TRIAL: NCT03741608
Title: A Mindfulness and Behavioral Intervention for Reducing Hypertension Among Women of Childbearing Age
Brief Title: B'More for a Peaceful Motherhood Hypertension Control Study
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID prevented us from continuing recruitment and interventions at community sites
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, Wendy Lane, Associate Professor, University of Maryland, Baltimore
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HP-00082822
Record Dates: First submitted 2018-11-12; First posted 2018-11-15 (Actual); Last update posted 2021-04-14 (Actual); Status verified 2021-04

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Intervention Model Description: Two groups will both participate in the 7-part educational series to reduce high blood pressure. One of the two groups will also be given a blood pressure cuff and will be trained to check their own blood pressure. We will track blood pressure and stress level of both groups for 6 months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Education, BP cuff & training (Active Comparator): High blood pressure management education. Home blood pressure measurement
  Interventions: Behavioral: High blood pressure management education; Behavioral: Home blood pressure measurement
- Education only (Active Comparator): High blood pressure management education
  Interventions: Behavioral: High blood pressure management education

INTERVENTIONS:
Behavioral: High blood pressure management education — The 7-part education series includes 5 sessions focused on mindfulness and breathing techniques for stress reduction. One session will focus on choosing healthy, low salt foods and will provide resources for smoking cessation. The final session will include a grocery store tour to teach participants how to read food labels and to purchase healthy food.
Behavioral: Home blood pressure measurement — Participants will be taught to use an automated blood pressure cuff and will be asked to provide monthly blood pressure readings to study staff.
  Arms: Education, BP cuff & training

SUMMARY:
This study will assess whether an intervention including mindfulness, dietary education, and smoking cessation can help African-American women of childbearing age (age 18-44) with hypertension or high blood pressure to lower their blood pressure. The investigators propose to screen women of childbearing age for hypertension, and to invite women to participate in an intervention to reduce their blood pressure. The investigators will track their perceived stress and their blood pressure levels over the next 6 months. Half of the women who participate will be given a blood pressure cuff and taught to measure their own blood pressure. More frequent tracking of blood pressure will be done in these women.

DETAILED DESCRIPTION:
Chronic and pregnancy-associated hypertension increase risk for poor birth outcomes, including higher rates of low birthweight and preterm birth. Mindfulness interventions, dietary education, and smoking cessation education have all been effectively employed to reduce hypertension, but have infrequently targeted women of childbearing age in community settings. This study will screen African-American women of childbearing age for hypertension, and invite women with hypertension to participate in a seven-session intervention to reduce blood pressure. The investigators will track their perceived stress and their blood pressure levels over the next 6 months. Half of the women who participate will be given a blood pressure cuff and taught to measure their own blood pressure. More frequent tracking of blood pressure will be done in these women.

ELIGIBILITY:
Inclusion Criteria:

* Hypertension
* Age 18-44
* African-American
* Female

Exclusion Criteria:

* Male
* Age <18 or >44
* Non-African American
* Not female
* Pregnant

Ages: 18 Years to 44 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — women
Enrollment: 23 (Actual)
Dates: Start 2019-01-22 (Actual); Primary Completion 2020-04-01 (Actual); Study Completion 2020-04-01 (Actual)

PRIMARY OUTCOMES:
Blood pressure reduction | 6 months
  decrease in systolic and diastolic blood pressure by 10 points each

SECONDARY OUTCOMES:
Stress | 6 months
  Score on Perceived Stress Scale. The Perceived Stress Scale (Cohen, S, 1994) is the most widely used psychological instrument for measuring the perception of stress. It is a 10-question survey asking to what degree certain stressors have been a problem in the past month. Responses are recorded on a 5-point Likert scale from 0 (never) to 4 (very often). The 6 negatively-stated items are scored as is, while the four positively stated items' scores are reversed. The total score may therefore range from 0 to 40. Higher scores indicate higher levels of stress (i.e. a worse outcome). There are no subscales.

CONTACTS AND LOCATIONS:
Overall Officials: Wendy G Lane, MD, MPH, Principal Investigator — University of Maryland, College Park
Locations (4):
- United States (4):
  - Leonard E. Hicks Community Center, Baltimore, Maryland
  - Furman L. Templeton Preparatory Academy, Baltimore, Maryland
  - Pedestal Gardens Apartment Homes, Baltimore, Maryland
  - Union Baptist Harvey Johnson Head Start Program, Baltimore, Maryland

IPD SHARING:
Plan to Share IPD: No
We will share blood pressure measurements and Perceived Stress Scale measurements upon request